CLINICAL TRIAL: NCT00829777
Title: A Phase-I, Two-Stage, Double-Blind, Placebo-Controlled, Pharmacokinetic and Pharmacodynamic Trial of Low Doses of Intravenous 6β-Naltrexol (AIKO-150) in Opioid-Dependent Subjects.
Brief Title: Safety Study of Intravenous 6β-Naltrexol (AIKO-150) in Opioid-Dependent Subjects
Acronym: AIKO-150
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Responsible Party: John Mendelson, M.D., Principal Investigator, Addiction & Pharmacology Research Laboratory, California Pacific Medical Center Research Institute
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 28.073-2; PR#0830A; IRB# 26.073-2
Record Dates: First submitted 2009-01-23; First posted 2009-01-27 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Opiate Addiction
Keywords: Naloxone; 6β-Naltrexol; Opioid-dependent; Pharmacokinetics; peripheral effects of withdrawal; central effects of withdrawal
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Naloxone; Lactulose

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 6β-Naltrexol escalating doses from 0.05-0.5 mg IV — Drug: Naloxone 0.1 mg IV/5 minutes to all subjects to determine tolerability to precipitated withdrawal during screening. Those that tolerate withdrawal proceed to Stage 1:
  Drug: Lactulose 10 gm orally plus 3 IV infusions 30 minutes apart of Naloxone 0.1 mg IV and 2 placebo given randomly to all subjects. If tolerated, proceed to 5 additional medication dosing sessions with all subjects receiving oral Lactulose 10 GM plus IV escalating 6β-Naltrexol 0.05 mg, 0.15 mg, 0.5 mg with a randomized placebo.
  Other Names: Naloxone; 6β-Naltrexol; Lactulose

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of intravenous 6β-Naltrexol administered to opiate dependent subjects

ELIGIBILITY:
Inclusion Criteria:

* Opiate dependent males and females age 21-45 on stable doses of methadone
* Fluent English speaker
* Willing and able to give written consent

Exclusion Criteria:

* Pregnancy or lactation

FOR MORE DETAILS CONTACT THE RESEARCH CLINIC.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
- 6β-Naltrexol will have 13 hr half-life. Plasma collected | -0-24 hrs post dose
- 6β-Naltrexol pharmacokinetic profile in opioid-dependent population will be similar in non-opioid-dependent population. Plasma levels collected | 0-8 hrs post dose

SECONDARY OUTCOMES:
-6β-Naltrexol will have a lower potency in precipitating withdrawal and be better tolerated than Naloxone assessed by vital signs, objective/subjective ate Withdrawal Scales, Visual Analog Scales, Pupil Size and GI Motility measures | 0-8 hrs post dose
6β-Naltrexol dose-dependent increases to reverse methadone-induced bowel dysfunction. Plasma levels and Hydrogen Breath Tests | 0-8 hrs post dose

CONTACTS AND LOCATIONS:
Overall Officials: John E Mendelson, MD, Principal Investigator — California Pacific Medical Center Research Institute
Locations (1):
- CPMC Addiction & Pharmacology Research Laboratory (APRL), San Francisco, California, United States